CLINICAL TRIAL: NCT02735629
Title: Antagonism of Opioid-Induced Respiratory Depression by CX1739 With Preservation of Opioid Analgesia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RespireRx (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CRTX-05
Record Dates: First submitted 2016-03-23; First posted 2016-04-13 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Opiate Induced Respiratory Depression
MeSH Terms: interventions — Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- CX1739 - 300 mg (Experimental): Study Drug - low dose
  Interventions: Drug: CX1739 - 300 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- CX1739 - 600 mg (Experimental): Study drug - mid Dose
  Interventions: Drug: CX1739 - 600 mg
- CX1739 - 900 mg (Experimental): Study drug - high dose
  Interventions: Drug: CX1739 - 900 mg

INTERVENTIONS:
Drug: CX1739 - 300 mg — Ampakine CX1739 - 300 mg
  Other Names: Low dose
  Arms: CX1739 - 300 mg
Drug: CX1739 - 600 mg — CX1739 - 600 mg
  Other Names: mid dose
  Arms: CX1739 - 600 mg
Drug: CX1739 - 900 mg — CX1739 - 900 mg
  Other Names: high dose
  Arms: CX1739 - 900 mg
Drug: Placebo — Placebo to 300 mg CX1739
  Other Names: Placebo to 300 mg CX1739
  Arms: Placebo

SUMMARY:
The study is an investigation to assess the capacity of ascending doses of CX1739 to antagonize the respiratory depressive effect of remifentanil. The study will also investigate whether ascending doses of CX1739 reduce the analgesic effect of remifentanil or alter the BIS measure of sedation and will evaluate the safety of CX1739 when used in conjunction with remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for this trial, subjects must meet all of the following criteria:

  1. Males 18 to 50 years of age, inclusive
  2. Body mass index of 18.0 to 30.0 kg/m2, inclusive, using the formula: weight (kg)/height (m)2
  3. Healthy, as determined by medical history, physical examination including vital signs, and clinical laboratory test results
  4. American Society of Anesthesiologists Physical Status Classification 1
  5. Willing and able to provide voluntary, written informed consent

Exclusion Criteria:

* If a subject meets any of the following criteria, he cannot be enrolled in the study:

  1. History of any chronic illness or evidence of clinically significant organic or psychiatric disease on medical history or physical examination which, in the opinion of the principal investigator (PI), would confound the study results or present a risk to the subject
  2. Acute illness within 2 weeks before dosing
  3. History of any clinically significant pulmonary condition (eg, asthma) within the last 2 years requiring admission to the hospital
  4. Previous diagnosis of obstructive sleep apnea based on polysomnography
  5. Currently using any prescription medication or use within the last 30 days
  6. Laboratory values (clinical chemistry, hematology, urinalysis) outside the laboratory reference range considered clinically significant (NOTE: in the event of any parameter lying outside of the normal range, the sample may be repeated once; this value will be accepted if it lies within the normal range)
  7. Presence of QT interval corrected > 440 msec on ECG
  8. Resting HR while awake < 45 or > 90 beats/minute
  9. History of daily use of tobacco or other nicotine-containing products within 1 year of study entry or positive cotinine test at screening and subsequent study visits
  10. History of allergic hypersensitivity to ampakines (CX717, CX1739), remifentanil, naloxone, or any component of these formulations; history of multiple drug allergies
  11. History or current evidence of abuse of any drug substance, licit or illicit, including alcohol; positive urine drug screen (UDS) for drugs of abuse at screening
  12. Inability to understand the protocol requirements; instructions; study-related restrictions; or nature, scope, and possible consequences of the study
  13. Unlikely to complete the study, eg, because of inability to return for follow-up visits
  14. Participation in another study with any investigational drug in the 3 months preceding this study
  15. Blood or plasma donation of more than 500 mL during the month before randomization and more than 50 mL in the 2 weeks before randomization

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Respiratory depression | Sequence #1 - 30 minutes
  Respiratory rate, tidal volume, minute volume as determined by plethysmography

SECONDARY OUTCOMES:
Pain tolerance threshold | Sequence #2 - 20 minutes
  Analgesia assessed by pain tolerance threshold to 5, 250, and 2000 Hertz sine-wave electrical stimulation using the quantitative sensory testing device - Neurometer
Maintenance of sedation | Sequence #1 - 30 minutes
  Bispectral index (BIS) measure of sedation
The number of patients that experience an adverse drug reaction upon ingestion of CX1739 when used alone or in conjunction with remifentanil | up to 5 weeks
  Vital signs, including noninvasive blood pressure, heart rate, RR, end-tidal carbon dioxide, pulse oximetry saturation, and temperature
  * Electrocardiograms
  * Focused physical examinations
  * Adverse events
Change in pupil size | Sequence #2 - 20 minutes
  Pupil size will be assessed intermittently with a noninvasive pupillometer incorporated into a pair of glasses placed on the subject's head

CONTACTS AND LOCATIONS:
Overall Officials: Richard Purcell, Study Director — RespireRx Pharmaceuticals
Locations (1):
- Duke Clinical Research Unit, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No